CLINICAL TRIAL: NCT03572894
Title: Comparison of PVI and RPVI During a Tidal Volume Challenge Under General Anesthesia: A Prospective Validation Pilot Study
Brief Title: Comparison of PVI and RPVI
Acronym: RPVI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0313
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-06

CONDITIONS: Venous; Return (Anomaly)
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PVI and RPVI measurements — PVI and RPVI measurements during variations of the tidal volume (Vt challenge) and a recruitment maneuver in anesthetized and mechanically ventilated patients.
  * T0 : Vt 6 mL/kg of predicted body weight (PBW) during 5 minutes
  * T1 : Vt 8 mL/Kg of PBW during 5 minutes
  * T2 : Vt 10 mL/kg of PBW during 5 minutes
  * T3 : Vt 6 mL/kg of PBW during 5 minutes
  * T4 : A single recruitment maneuver
  Data will be recorded at each step.

SUMMARY:
Pleth Variability Index (PVI) is a non-invasive and automated measure of the respiratory variations of plethysmography during mechanical ventilation. PVI is extracted via an algorithm implemented on Masimo Radical 7 device (Masimo, Irvine, CA). PVI is commonly used in anesthesiology and has been validated to predict fluid responsiveness and optimize fluid administration in the surgical setting. However, the signal/noise ratio of PVI makes acute changes in PVI somewhat difficult to interpret at the bedside. Subsequently, a new algorithm entitled RPVI (Rainbow Pleth Variability Index), has been developed in order to improve the signal/noise ratio of PVI and facilitate its clinical use by practitioners. The details of this new proprietary built-in algorithm are unknown and no data are available to date. Therefore, the main objective of the study was to compare RPVI and PVI during dynamic changes in venous return induced by a tidal volume (Vt) challenge during mechanical ventilation in anesthetized patients. The hypothesis was that the agreement between both dynamic indices would be good.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Low or intermediate risk surgery or noninvasive procedures in the supine position
* General anaesthesia and volume-controlled mechanical ventilation.

Exclusion Criteria:

* Non sinus heart rhythm
* Left Ventricular Ejection Fraction < 50%
* Documented right ventricle failure
* Lack of patient consent
* Pregnancy
* Minor patient or under tutorship
* Presence of spontaneous ventilatory movements (attested by a real respiratory rate higher than the set respiratory rate)
* Report HR / RR <3.6 (HR: heart rate, RR: respiratory rate)
* Open chest surgery
* Laparoscopic surgery
* Vital or lateral decubitus surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing closed-chest surgery in the supine position under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnostic characteristics of RPVI in comparison to PVI | 30 minutes
  Agreement and interchangeability of RPVI and PVI: Bland Altman analysis for repeated measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation, Hôpital Cardiologique Louis Pradel, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No